CLINICAL TRIAL: NCT05311787
Title: The Strategy of Implementation of the ERAS Protocol After Esophageal Surgery Based on Innovative Technologies
Brief Title: The Strategy of Implementation of the ERAS Protocol After Esophageal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vishnevsky Center of Surgery (Other)
Responsible Party: Principal Investigator, Maria Yan, Principal Investigator, Vishnevsky Center of Surgery
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 315030310071
Record Dates: First submitted 2022-03-22; First posted 2022-04-05 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: ERAS; Esophageal Diseases
MeSH Terms: conditions — Esophageal Diseases | interventions — Esophagectomy

STUDY DESIGN:
Intervention Model Description: All the patients over 18 years old with esophageal diseases who are required surgical treatment include in trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early oral feeding (Other): The part of our investigation was prostective randomised trial which compared the result of patients with early oral feeding (since first day) and traditional group (oral feeding since 5th day)
  Interventions: Procedure: esophagectomy with simultaneous reconstruction

INTERVENTIONS:
Procedure: esophagectomy with simultaneous reconstruction — Subtotal resection of esophagus and simultaneous reconstruction by gastric pull-up or colon conduit
  Other Names: esophagectomy with gastric pull-up; esophagectomy with colon conduit; McKeown; transhiatal esophagectomy

SUMMARY:
Application of the perioperative enhanced recovery protocol has allowed to carry out esophagectomy to the patients with severe comorbidities and has led reducing the risks of severe postoperative complications.

DETAILED DESCRIPTION:
The clinical trial included the parients who participated in the protocol ERAS since 2011, who uderwent esophagectomy with simultaneous reconstruction. The parients had benign or malignant esophageal diseases. The ERAS protocol consisted of components of perioperative recovery. The number of patients until now has reached 400 patients. During trial there was modifications of aspects of ERAS protocol such as a rejection of nasogastric tube or cervical drenage. The role of multidisplinary team is the main success of the result of the implemented ERAS protocol.

ELIGIBILITY:
Inclusion Criteria:

* all patients with esophageal diseases

Exclusion Criteria:

* before 18 years old
* who do not need surgery as a treatment
* who not underwent simultaneous recontruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
mortality | 30 days
  the rate of mortality after surgery
morbidity | 30 days
  the rate of morbidity after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mary Yan, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
all IPD
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: By the 2026, open access

REFERENCES:
- See also: Related Info — https://intensive-care.ru/rannee-peroralnoe-pitanie-kak-komponent-programmy-uskorennogo-vosstanovleniya-posle-subtotalnoj-ezofagektomii-s-odnomomentnoj-plastikoj-pishhevoda-prospektivnoe-randomizirovannoe-issledovanie/